CLINICAL TRIAL: NCT03824977
Title: Prognostic Value of the 6-minute Stepper Test in Non-small Cell Lung Cancer Surgery
Acronym: PREOTEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02694-51
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Lung Neoplasm Malignant; Resectable Lung Non-Small Cell Carcinoma
Keywords: lung resection; low technology; six minutes stepper test; sit to stand test; physiotherapy; lung surgery; post-operative complications
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Six minutes stepper test (6MST) — The 6MST is done using a stepper (Stepper essential, Decathlon(TM), France), with a walking height of 20 cm, placed in front of a wall or parallel bars, so patients can hold on if necessary.
  Patients are instructed to make the maximum number of steps possible in 6 minutes, and are given a time check at one minute intervals.
Diagnostic Test: Sit to stand test (STST) — The STST is done using a chair measuring 47 cm in height. The patient are instructed to sit in the chair and then to do the maximum number of lifts possible from the chair, in 1 minute, with arms folded and without leaning against the chair.

SUMMARY:
The objective of this study is to evaluate the performances of the Six-Minute Stepper Test (6MST) and Sit To Stand test (STST) to predict post-operative complications after minimally invasive lung cancer resection.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Non-small cell lung cancer stage I to II, justifying major resection by VATS or RATS (segmentectomy, lobectomy, pneumonectomy), with or without histological confirmation

Exclusion Criteria:

* Partial or total amputation localized to the lower limb;
* Weight greater than 100 kg;
* Orthopedic, vascular or neurological disorders leading to the incapacity of realize the 6MST;
* Patient under tutorship or curatorship;
* Pregnant woman.
* Surgery canceled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients are included. On the day of the surgical consultation, the patient is informed of the modalities of the study by the thoracic surgeon and collects his non-opposition of participation. He is also evaluated by a physiotherapist, who supervises the realization of 6MST and STST.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
occurrence of a post-operative complication grade ≥ 2 on the Clavien-Dindo scale within three months after surgery | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Boujibar , F, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boujibar F, Gillibert A, Bonnevie T, Rinieri P, Montagne F, Selim J, Cuvelier A, Gravier FE, Baste JM. The 6-minute stepper test and the sit-to-stand test predict complications after major pulmonary resection via minimally invasive surgery: a prospective inception cohort study. J Physiother. 2022 Apr;68(2):130-135. doi: 10.1016/j.jphys.2022.03.001. Epub 2022 Apr 5. PMID 35396177